CLINICAL TRIAL: NCT02003430
Title: Functional Assessment and Radiation Adherence/Toxicity in Older and Younger Patients With Non-Ovarian Gynecological Cancers
Brief Title: Radiation Adherence/Toxicity in Patients With Non-Ovarian Gynecological Cancers
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1321
Record Dates: First submitted 2013-11-18; First posted 2013-12-06 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Non-ovarian Gynecological Cancers
Keywords: gynecologic malignancy; non-ovarian gynecological cancer; cervical cancer; vaginal cancer; vulvar cancer; endometrial cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ≥65 years old: 20 patients greater than or equal to 65 years of age
- <65 years old: 20 patients less than 65 years of age

SUMMARY:
The purpose of this study is to investigate the association between the Independent Activities of Daily Living (I-ADL) component of the Comprehensive Geriatric Assessment (CGA) and poor tolerance to radiation treatment in older and younger patients with non-ovarian gynecological cancers.

DETAILED DESCRIPTION:
There are little data regarding the impact of functional age on tolerance to radiotherapy for gynecologic cancers. A comprehensive geriatric assessment (CGA) tool which measures functional status (including the Instrumental Activities of Daily Living (I-ADL)), among many other important geriatric related conditions, was developed by Hurria and colleagues. Geriatric assessment variables including functional status predicted for toxicity in older patients receiving chemotherapy and surgery for multiple cancer types., 2 We hypothesize that I-ADL can be used to predict treatment tolerance in patients of all ages receiving pelvic and/or paraaortic region radiation therapy for gynecologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* ≥Age 18 years (no upper age limit)
* Diagnosis of cervical, vaginal, vulvar, or endometrial cancer with either pelvic radiotherapy or chemoradiotherapy planned as part of standard treatment.
* Consented for receipt of External Beam Radiation Therapy (EBRT) at the University of North Carolina Chapel Hill
* Ability to read English (required for CGA)
* Curative treatment intent as defined by their radiation oncologist
* Negative serum pregnancy test in women of childbearing potential

Exclusion Criteria:

* < Age 18 years
* Incurable cancer as defined by their radiation oncologist
* Planned radiation for palliative intent only
* Inability to complete the I-ADL section of the CGA
* Prior radiation to areas targeted by radiotherapy within this study
* Other active, invasive malignancy requiring active ongoing therapy during their radiotherapy with the exception of:
* Localized squamous cell carcinoma of the skin
* Basal-cell carcinoma of the skin
* Other malignancies requiring locally ablative therapy only

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 18 years of age or above with a diagnosis of cervical, vaginal, vulvar, or endometrial cancer with either pelvic radiotherapy or chemoradiotherapy planned as part of standard treatment with curative intent at the Department of Radiation Oncology at UNC Chapel Hill.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Pre-treatment I-ADL dependency | Pre-treatment
  Pre-treatment I-ADL dependency is defined as scoring less than 14 on the I-ADL scale of the CGA.

SECONDARY OUTCOMES:
Poor adherence to treatment | During or 4-8 weeks post-treatment
  Poor adherence to treatment is defined by at least one of the following:
  1. > 3 day treatment delay secondary to treatment related toxicity during radiation therapy.
  2. Hospitalization secondary to treatment related toxicity during or up to 4-8 weeks post radiation therapy.
  3. Unplanned dose reductions in either radiation or concurrent chemotherapy secondary to treatment related toxicity during radiation therapy
  4. Unplanned change in concurrent chemotherapy regimen secondary to treatment related toxicity during radiation therapy.

OTHER OUTCOMES:
Patient-reported acute grade 3-5 radiation related toxicities | During treatment and 4-8 weeks post-treatment
  Patient-reported acute grade 3-5 radiation related toxicities will be based on the PRO-CTCAE questionnaire during and 4-8 weeks post radiation therapy and at 6 months.
Provider-reported grade 3-5 acute radiation related toxicities | During treatment and 4-8 weeks post-treatment
  Provider-reported grade 3-5 acute radiation related toxicities will be based on the CTCAE (Common Toxicity Criteria for Adverse Effects) v4.03 during and 4-8 weeks post radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Varia, MD, ChB, Principal Investigator — Department of Radiation Oncology, University of North Carolina Chapel Hill; Noam VanderWalde, MD, Study Director — Department of Radiation Oncology, Unverisity of North Carolina Chapel Hill
Locations (1):
- UNC Department of Radiation Oncology Clinic, Chapel Hill, North Carolina, United States